CLINICAL TRIAL: NCT03895047
Title: Multifocal Tomographic Neurofeedback for Treating Chronic Tinnitus in Older People
Brief Title: ICCAC-ToNF & Tinnitus
Acronym: ICCAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-01035
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- dACC,I,AC (Active Comparator): Within each training session, participants will receive 7 minutes training for each of the three brain areas Insula (I), dorsal anterior cingulate cortex (dACC) & the auditory cortex (AC) resulting in 21Minutes of training for each session. The arm Title describes the order in which participants within this Arm will receive the three trainings. (E.g. dACC,I,AC: each participant in this group receives the training of the dACC first and the AC last.) This sequence order is kept stable during all training sessions.
  12 sessions of Neurofeedback Training, 1-2 times per week.
  Interventions: Other: tomographic EEG Neurofeedback Training
- dACC,AC,I (Active Comparator): Within each training session, participants will receive 7 minutes training for each of the three brain areas Insula (I), dorsal anterior cingulate cortex (dACC) & the auditory cortex (AC) resulting in 21Minutes of training for each session. The arm Title describes the order in which participants within this Arm will receive the three trainings. (E.g. dACC,I,AC: each participant in this group receives the training of the dACC first and the AC last.) This sequence order is kept stable during all training sessions.
  12 sessions of Neurofeedback Training, 1-2 times per week.12 sessions of Neurofeedback Training, 1-2 times per week.
  Interventions: Other: tomographic EEG Neurofeedback Training
- I,dACC,AC (Active Comparator): Within each training session, participants will receive 7 minutes training for each of the three brain areas Insula (I), dorsal anterior cingulate cortex (dACC) & the auditory cortex (AC) resulting in 21Minutes of training for each session. The arm Title describes the order in which participants within this Arm will receive the three trainings. (E.g. dACC,I,AC: each participant in this group receives the training of the dACC first and the AC last.) This sequence order is kept stable during all training sessions.
  12 sessions of Neurofeedback Training, 1-2 times per week.
  Interventions: Other: tomographic EEG Neurofeedback Training
- I,AC,dACC (Active Comparator): Within each training session, participants will receive 7 minutes training for each of the three brain areas Insula (I), dorsal anterior cingulate cortex (dACC) & the auditory cortex (AC) resulting in 21Minutes of training for each session. The arm Title describes the order in which participants within this Arm will receive the three trainings. (E.g. dACC,I,AC: each participant in this group receives the training of the dACC first and the AC last.) This sequence order is kept stable during all training sessions.
  12 sessions of Neurofeedback Training, 1-2 times per week.
  Interventions: Other: tomographic EEG Neurofeedback Training
- AC,dACC,I (Active Comparator): Within each training session, participants will receive 7 minutes training for each of the three brain areas Insula (I), dorsal anterior cingulate cortex (dACC) & the auditory cortex (AC) resulting in 21Minutes of training for each session. The arm Title describes the order in which participants within this Arm will receive the three trainings. (E.g. dACC,I,AC: each participant in this group receives the training of the dACC first and the AC last.) This sequence order is kept stable during all training sessions.
  12 sessions of Neurofeedback Training, 1-2 times per week.
  Interventions: Other: tomographic EEG Neurofeedback Training
- AC,I,dACC (Active Comparator): Within each training session, participants will receive 7 minutes training for each of the three brain areas Insula (I), dorsal anterior cingulate cortex (dACC) & the auditory cortex (AC) resulting in 21Minutes of training for each session. The arm Title describes the order in which participants within this Arm will receive the three trainings. (E.g. dACC,I,AC: each participant in this group receives the training of the dACC first and the AC last.) This sequence order is kept stable during all training sessions.
  12 sessions of Neurofeedback Training, 1-2 times per week.
  Interventions: Other: tomographic EEG Neurofeedback Training

INTERVENTIONS:
Other: tomographic EEG Neurofeedback Training — EEG-Electrodes are placed on the patients head to record the brain activity, EEG-recordings are processed by the standardized Low Resolution Brain Electromagnetic Tomography algorithm (sLORETA) to calculate the frequency spectrum in the auditory cortex, the insula and the anterior cingulate cortex and deliver feedback for the patient

SUMMARY:
Prevalence of chronic subjective tinnitus is rising with age and associated with maladaptive oscillatory changes in auditory as well as non-auditory regions of the brain such as the insula and the anterior cingulate cortex which are known to be key points within the salience and distress networks of the brain.Thus, we are conducting a clinical trial by implementing those auditory as well as non-auditory regions into a tomographical neurofeedback Training (ToNF) -protocol.

Prior to 12 electroencephalography (EEG) -based ToNF-trainings with 36 older participants using standardized Low Resolution Electromagnetic Tomography Software (sLORETA, Pascual-Marqui 2002), participants' brains will be measured using structural magnet resonance imaging (sMRI) in order to identify potential structural markers for training success (e.g. cortical thickness).

Training success will be measured by oscillatory change via EEG before and after the training period as well as by means of follow-up measures. Furthermore, a comprehensive battery of behavioral and psychometric standardized self-report questionnaires will be applied.

Based on this multifocal (Insula, dorsal anterior cingulate cortex & auditory cortex) ToNF we expect oscillatory changes resulting in decreased tinnitus symptoms such as perceived loudness and distress.

ELIGIBILITY:
Inclusion Criteria:

* chronic tinnitus (>6 months)
* Age 40 to 80
* Informed Consent
* Fluent in German language
* mentally & physically fit

Exclusion Criteria:

* ferromagnetic implants
* cochlear implants
* average hearing loss over 50 dB
* claustrophoby
* addiction to alcohol or drugs
* intake of anesthetics, tranquilizers, neuroleptics or antiepileptics
* acute suicidal

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tinnitus symptoms assessed by questionnaires | Time Frame: at 1, 3, 6 month follow up
  Assessement of the Tinnitus symptoms before and after the Treatment with neurofeedback by different questionnaires
Change from Baseline in frequency band EEG-activity in the auditory cortex, insula & dorsal anterior cingulate cortex | Time Frame: at 1, 3, 6 month follow up
  EEG recordings of the trained frequency bands are compared before and after the Intervention in the named time periods

SECONDARY OUTCOMES:
brain structure (volume, surface area) of the three regions of interest as predictor for training success. | Baseline (measurement before training)
  MRI measurement before training

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Division of Otorhinolaryngology ORL, Zurich, Canton of Zurich, Switzerland